CLINICAL TRIAL: NCT01913886
Title: Autologous Grafting of Mesenchymal Stem Cells in Severe Refractory Ischemic Cardiomyopathy
Brief Title: Mesenchymal Stem Cells to Treat Ischemic Cardiomyopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandra Cristina Senegaglia (Other)
Collaborators: Santa Casa de Misericórdia de Curitiba, Brazil (Unknown); Fundação Araucária (Other)
Responsible Party: Sponsor-Investigator, Alexandra Cristina Senegaglia, PhD, Pontifícia Universidade Católica do Paraná
Organization: Pontifícia Universidade Católica do Paraná (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC_Isquemica
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2016-09

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Cardiovascular Diseases; Myocardial Ischemia; Coronary Artery Disease; Heart Diseases; Coronary Disease; Ventricular Dysfunction; Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia; Coronary Artery Disease; Heart Diseases; Coronary Disease; Ventricular Dysfunction; Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSCs injection (Experimental): Injection of autologous bone marrow-derived mesenchymal cells
  Interventions: Procedure: MSCs injection

INTERVENTIONS:
Procedure: MSCs injection — MSCs cells will be injected in two aliquots of 10 ml by catheterism

SUMMARY:
This study will evaluate the safety and efficacy of intracoronary injection of mesenchymal stem cells (MSCs) to repair heart function in patients with myocardial ischemia.

DETAILED DESCRIPTION:
Ischemic heart disease is a major public health problem in the industrialized and developing world. Current research is focusing on the development of cell-based therapies using stem cells to treat heart failure. Mesenchymal stem cells (MSCs) can differentiate into endothelial cells and participate in the development of new blood vessels in the heart damaged. Therefore, MSCs has shown promise for heart repair. The investigators study will evaluate the safety and efficacy of intracoronary injection of mesenchymal stem cells (MSCs) to repair heart function in patients with myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary artery disease
* NYHA (Heart failure) Class II-IV or Angina pectoris CCS Class III or IV or symptoms consistent with.
* Ejection fraction between 35% and 55%.
* Stable medical therapy for at least one month
* Patients clinically treated with coronary angioplasty with or without intraluminal stent.
* Patients with surgical revascularization and without the possibility of new invasive intervention.

Exclusion Criteria:

* Human immunodeficiency virus (HIV1-2), HTLV-1 and 2.
* An active uncontrolled infection.
* Pregnancy.
* Mental disability.
* Terminal illnesses.
* Valvular heart disease, congenital heart disease or other causes of cardiomyopathy than ischemic.
* Life perspective by other diseases under 1 year.
* History of severe arrhythmias
* Renal dysfunction or against medication
* Inability to perform cardiac catheterization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in left ventricular ejection fraction (LVEF) measured by echocardiogram. | 3 months

SECONDARY OUTCOMES:
Change in quality of life | 3 months, 6 months, 12 months
  Measures by specific questionnaire of quality of life: Minnesota Living with Heart Failure Questionnaire (MLHFQ)
Changes in exercise capacity | 1 year
Changes in plasma inflammatory markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Brofman, PhD, Principal Investigator — Pontifícia Universidade Católica do Paraná
Locations (1):
- Pontifícia Universidade Católica do Paraná, Curitiba, Paraná, Brazil